CLINICAL TRIAL: NCT00315770
Title: Health of Young European Families and Fish Consumption
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Landspitali University Hospital (Other)
Collaborators: European Commission (Other); University of Iceland (Other); University College Cork (Other); University of Navarra (Other); The National Research Institute on Agriculture and Fisheries Research, Lisbon, Portugal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FQS-506359
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Overweight; Metabolic Syndrome X; Bone Resorption
Keywords: overweight; Metabolic syndrome
MeSH Terms: conditions — Overweight; Metabolic Syndrome; Bone Resorption | interventions — Diet, Reducing

INTERVENTIONS:
Procedure: weight loss diets for young adults

SUMMARY:
This is a controlled, randomized, intervention trial (CRIT) with 20-40 year old overweight individuals (n = 320) across Europe in order to distinguish between biologically active components of seafood, i.e., seafood proteins and n-3 lipids, regarding their effects on risk factors for metabolic syndrome, bone health, and weight management.

DETAILED DESCRIPTION:
Subjects were recruited through advertisements from October 2004 until April 2005. Recruitment of 320 subjects (140 from Iceland, 120 from Spain, and 60 from Ireland). The inclusion criteria were body mass index (BMI) 27.5 to 32.5 kg/m2, age 20-40 years, and a waist circumference of equal or more than 94 cm and 80 cm for men and women, respectively. Exclusion criteria were weight change due to weight loss diet within 3 months before the start of the study, use of supplements giving n-3 fatty acids, calcium or vitamin-D during the last three months, drug treatment of diabetes mellitus, hypertension or hyperlipidemia and women's pregnancy or lactation. Each subject was instructed to follow a diet, energy-restricted by 30% from estimated energy expenditure (approximately 600 kcal/day), for 8 consecutive weeks. The subjects were randomly assigned to four diets varying in types of dietary protein and amount of n-3 fatty acids (especially very long chain n-3 fatty acids):

I: no seafood (control, including 6 placebo capsules/day)

II: lean fish (150 g cod x 3/week)

III: fatty fish (150 g salmon x 3/week)

IV: fish-oil capsules (6 capsules/day)

Risk factors for metabolic syndrome, bone health and weight management were analysed at baseline and endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 27.5 to 32.5 kg/m2
* Ages 20-40 years
* Waist circumference of equal or more than 94 cm and 80 cm for men and women, respectively

Exclusion Criteria:

* Weight change due to weight loss diet within 3 months before the start of the study
* Use of supplements giving n-3 fatty acids
* Calcium or vitamin D during the last three months
* Drug treatment for diabetes mellitus
* Hypertension or hyperlipidemia
* Women's pregnancy or lactation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320
Dates: Start 2004-01; Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Weight loss
Anthropometry

SECONDARY OUTCOMES:
Blood lipid profile (total high-density lipoprotein [HDL]- and low-density lipoprotein (LDL)-cholesterol, triacylglycerol)
Fatty acid composition of red blood cells
Fasting plasma glucose and fasting insulin
C-reactive protein
Prostaglandins
Interleukins
Intercellular adhesion molecules
Vascular cell adhesion molecules
Antioxidants/pro-oxidants
Serum ghrelin
Leptin
Quantitative insulin-sensitivity check index (QUICKI)
Adiponectin
Plasminogen activator inhibitor (PAI-1)
Cortisol
Glutathione (GSH) reductase
Malondialdehyde
Bone specific alkaline phosphatase
Osteocalcin
Parathyroid hormone (PTH)
25-hydroxyvitamin D3 [25(OH) D3]
Creatinine
Pyridinoline (Pyr) and deoxypyridinoline (Dpyr)
Visual analogue scale for satiety

CONTACTS AND LOCATIONS:
Overall Officials: Inga Thorsdottir, PhD, Principal Investigator — LSH & HI

REFERENCES:
- [Derived] Ramel A, Halldorsson TI, Tryggvadottir EA, Martinez JA, Kiely M, Bandarra NM, Thorsdottir I. Relationship between BMI and body fatness in three European countries. Eur J Clin Nutr. 2013 Mar;67(3):254-8. doi: 10.1038/ejcn.2013.6. Epub 2013 Jan 30. PMID 23361157
- [Derived] Ramel A, Martinez JA, Kiely M, Bandarra NM, Thorsdottir I. Effects of weight loss and seafood consumption on inflammation parameters in young, overweight and obese European men and women during 8 weeks of energy restriction. Eur J Clin Nutr. 2010 Sep;64(9):987-93. doi: 10.1038/ejcn.2010.99. Epub 2010 Jun 16. PMID 20551965
- [Derived] Ramel A, Martinez JA, Kiely M, Bandarra NM, Thorsdottir I. Moderate consumption of fatty fish reduces diastolic blood pressure in overweight and obese European young adults during energy restriction. Nutrition. 2010 Feb;26(2):168-74. doi: 10.1016/j.nut.2009.04.002. Epub 2009 May 31. PMID 19487105
- [Derived] Ramel A, Parra D, Martinez JA, Kiely M, Thorsdottir I. Effects of seafood consumption and weight loss on fasting leptin and ghrelin concentrations in overweight and obese European young adults. Eur J Nutr. 2009 Mar;48(2):107-14. doi: 10.1007/s00394-008-0769-9. Epub 2009 Jan 13. PMID 19142567
- [Derived] Ramel A, Martinez A, Kiely M, Morais G, Bandarra NM, Thorsdottir I. Beneficial effects of long-chain n-3 fatty acids included in an energy-restricted diet on insulin resistance in overweight and obese European young adults. Diabetologia. 2008 Jul;51(7):1261-8. doi: 10.1007/s00125-008-1035-7. Epub 2008 May 20. PMID 18491071
- [Derived] Lucey AJ, Paschos GK, Cashman KD, Martinez JA, Thorsdottir I, Kiely M. Influence of moderate energy restriction and seafood consumption on bone turnover in overweight young adults. Am J Clin Nutr. 2008 Apr;87(4):1045-52. doi: 10.1093/ajcn/87.4.1045. PMID 18400730